CLINICAL TRIAL: NCT01446588
Title: Ocular Hypertension And Yoga Study
Acronym: OHAYS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No Funding was acquired.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Pamela Jeter, Postdoctoral Research Fellow, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00041019
Record Dates: First submitted 2011-09-20; First posted 2011-10-05 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Ocular Hypertension; Sleep Disturbance; Stress; Anxiety; Depression
MeSH Terms: conditions — Ocular Hypertension; Parasomnias; Anxiety Disorders; Depression | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Yoga (Experimental): Yoga group
  Interventions: Behavioral: Yoga Intervention

INTERVENTIONS:
Behavioral: Yoga Intervention — Three yoga classes per week for 8 weeks.
  Other Names: Yoga, Ashtanga

SUMMARY:
The investigators aim to pilot test the efficacy of a yoga intervention designed specifically for individuals with ocular hypertension. The investigators would like to find out if a combination of breathing, postures and meditation may help to reduce intraocular pressure in the short term after each yoga session, and also long-term across an 8-week program. Subjects will participate in the yoga intervention sessions led by Dr. Pamela Jeter once a week at the investigators center, and will be asked to practice at home at least twice a week using a audio CD.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Diagnosis of ocular hypertension not requiring treatment of IOP
* IOP in at least one eye ≥ 21 mm Hg
* Normal Humphrey 24-2 or 30-2 visual fields for both eyes as determined by the patient's glaucoma specialist
* Best-corrected visual acuity better than 20/40 in both eyes
* Being healthy to the extent that participation in yoga therapy would not exacerbate any existing disease conditions;
* Participants do not engage in athletic activity on a regular basis (i.e. are sedentary)
* Able and willing to participate on a weekly basis for the 11-week intervention;
* Informed consent

Exclusion Criteria:

VISUAL HISTORY

* Any visual field loss in either eye consistently detected with Humphrey Visual Field 30-2 or 24-2
* Inability to understand study procedures or communicate responses to visual stimuli in a consistent manner (cognitive impairment)
* Previous intraocular surgery, except for uncomplicated extracapsular cataract extraction with posterior chamber-intraocular lens implant and no escape of vitreous to the anterior chamber, strabismus, cosmetic eyelid surgery, and radial keratotomy
* Secondary causes of elevated IOP, including ocular and systemic corticosteroid use
* Angle closure glaucoma or anatomically narrow angles-75% of the circumference of the angle must be grade 2 or more by Shaffer criteria
* Pigmentary glaucoma
* Congenital glaucoma
* Other diseases that cause visual field loss or optic disc abnormalities
* Difference in cup-disc ratios (horizontal by contour) between the two eyes of >0.2
* Background diabetic retinopathy, defined as at least 1 microaneurysm seen on ophthalmoscopy with dilated pupil, or any retinal hemorrhage

SPECIFIC SYSTEMIC DISEASES/CONDITIONS

* Abdominal Aneurism
* Cancer, metastatic
* Fibromyalgia, severe
* Inflammatory autoimmune diseases (e.g. Lupus, Rheumatoid arthritis, Scleroderma)
* Other disabling chronic conditions (e.g., disabling heart or lung disease, diabetic neuropathy, receiving treatment for hepatitis)
* A life-threatening or debilitating disease

BACK PROBLEM OF COMPLICATED NATURE, INCLUDING MEDICO-LEGAL ISSUES

* Seeking/receiving compensation/litigation for back pain
* Previous back surgery, ever
* Low back pain that has lasted > 1 month
* Severe pain when bending or twisting spine
* Sciatica
* Discitis or Disk disease
* Fracture of vertebra
* Infectious cause of back pain
* Scoliosis, severe or progressive
* Spinal stenosis
* Spondylolisthesis
* Anklyosing spondylitis

CONDITIONS THAT MIGHT MAKE IT DIFFICULT TO ATTEND THE CLASSES OR PRACTICE AT HOME.

* Deafness or severe hearing problems
* Psychoses, major
* Schedules do not permit participation in classes or home practice (including planning to move out of town)
* Paralysis
* Unable to walk two city blocks
* Unable to get up and down from floor
* Lack of transportation
* Any planned surgery during the upcoming study period

CONDITIONS/CIRCUMSTANCES THAT MIGHT CONFOUND TREATMENT EFFECTS OR INTERPRETATION OF DATA

* Pregnant or nursing women as determined by patient self-report
* Use of psychotropic medication
* Consumption of more than three alcoholic beverages per day
* Smoking more than 10 cigarettes per day
* Recent substance abuse

CONDITION WOULD MAKE IT DIFFICULT TO PROVIDE FULLY INFORMED CONSENT

* Dementia
* Long or short-term memory loss
* Unable to read or speak English

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure (IOP) | Change in IOP from mean baseline at 8-weeks (end of yoga intervention period)
  Baseline IOP measures will be obtained at two visits prior to the intervention. At each weekly visit, we will obtain two series of IOP measures about one hour apart, similar to the sequence that will be used during the weekly yoga intervention, to estimate trends over an 8-week intervention period. Post-intervention IOP will be measured at a single session one week after the yoga intervention has ended, and at a follow-up visit one month after the yoga intervention. Subjects will be masked to the IOP results until they have completed the study.

SECONDARY OUTCOMES:
Body Mass Index (BMI) (i.e. weight and height) | Week 0 and week 8
  Weight and height will be taken at baseline and Post-intervention.
Blood pressure | once a week for a total period of 11 weeks; then one additional measure 1 month later
  Systemic blood pressure (using a digital monitor with an automated cuff) and pulse rate will be measured at baseline, at the beginning and end of each yoga class, and the two post-intervention visits.
Respiratory Rate (RR) | Week 0 and Week 8
  Respiratory rate will be measured twice for each participant to reduce within-session variability. It will be determined by counting the number of inhalations with a stethoscope for 30 seconds at rest and multiplying by two at baseline and post-intervention.
Pittsburgh Sleep Quality Index (PSQI) | Week 0 and Week 8
  The 19-item PSQI questionnaire will be used to gauge sleep quality over the past month. It includes both qualitative and quantitative aspects of sleep, and evaluates seven subscale dimensions of sleep quality. Measured at baseline (week 0) and immediately after the 8-week intervention.
Perceived Stress Scale (PSS) | Week 0 and Week 8
  In order to subjectively assess the degree to which respondents have appraised situations in their life to be stressful on a given day, we will administer the 14 item PSS.
Beck Anxiety Index (BAI) | Week 0 and Week 8
  The 21 item BAI will be used to measure the severity of an individual's anxiety over the past month.
Beck Depression Index (BDI) | Week 0 and Week 8
  We will use the BDI to provide a measure of severity and type of depression.
Positive and Negative Affect Schedule (PANAS) | Week 0 and Week 8
  The PANAS questionnaire consists of 10 positive affect items, which reflect one's level of pleasurable engagement with the environment, and 10 negative affect items, which are a general factor of subjective distress.
Vision Test/Ocular Disease Catastrophizing Scale | Week 0 and Week 8
  The Catastrophizing Scale includes 20 questions that measure the individual's state and/or trait immediately after vision tests are performed.
Philadelphia Mindfulness Scale (PHLMS) | Week 0, Week 4 and Week 8
  This 20-item scale assesses two components of mindfulness, acceptance and awareness. Total scores on both subscales range from 20 to 100, higher scores reflect greater mindfulness. The PHLMS will be collected at baseline, during week 4 and post- intervention.
Exit Survey | Week 8
  Participants will complete a brief survey regarding their experience with the yoga class. The survey is comprised of open-ended and multiple-choice response items (e.g. treatment expectations).
Practice Log | once a week for a total period of 8 weeks
  Participants will be asked to complete a weekly log online to report the activity performed, time allotted to the practice and will be used to evaluate compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Ava Bittner, OD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Lions Vision and Research Rehabilitation, Baltimore, Maryland, United States